CLINICAL TRIAL: NCT04221126
Title: Thermo-mechanical Fractional Injury Enhances Skin Surface- and Epidermal- Protoporphyrin IX Fluorescence: Comparison of 5-aminolevulinic Acid in Cream and Gel Vehicles
Brief Title: TMFI Enhances Skin Surface and Epidermal PpIX Fluorescence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merete Haedersdal (Other)
Responsible Party: Sponsor-Investigator, Merete Haedersdal, PhD, Dr. med, Professor, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-004397-96
Record Dates: First submitted 2019-12-27; First posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Normal Skin
Keywords: protoporphyrin ix; 5-aminolevulinic acid; thermo-mechanical intervention; normal skin

STUDY DESIGN:
Masking Description: Randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- TMFI +cream (Experimental): TMFI + ALA cream
  Interventions: Device: TMFI; Drug: ALA cream
- TMFI + gel (Experimental): TMFI + ALA gel
  Interventions: Device: TMFI; Drug: ALA gel
- ALA creAM (Active Comparator): ALA cream
  Interventions: Drug: ALA cream
- ALA GEL (Active Comparator): ALA gel
  Interventions: Drug: ALA gel
- Control (No Intervention): Untreated control with no intervention

INTERVENTIONS:
Device: TMFI — Tixel rapidly transfer thermal energy by a metallic pyramid tip that enable skin contact through integrated pulsed movements. The rapid heating dehydrates he epidermis and superficial dermis and creates micropores with no coagulative damage of surronding tissue.
  Other Names: Thermo-mechanical fractional injury
  Arms: TMFI + gel; TMFI +cream
Drug: ALA cream — ALA compounded in a cream
  Other Names: 5-aminolevulinic acid compounded in a cream
  Arms: ALA creAM; TMFI +cream
Drug: ALA gel — ALA compounded in a gel
  Other Names: 5-aminolevulinic acid compounded in a gel
  Arms: ALA GEL; TMFI + gel

SUMMARY:
This study investigates a relatively new device TMFI and incubation of ALA in a cream-vehicle and a gel-vehicle.

DETAILED DESCRIPTION:
Topical photodynamic therapy (PDT) is a well-established treatment for dermatological pre-malignant actinic keratoses and Morbus Bowen as well as selected cases of basal cell carcinomas. PDT is exceedingly well suited for treatment of larger skin areas and provide excellent cosmetic results. PDT is based on the photosensitizing drug 5-aminolevulinic acid (5-ALA) that is metabolized into the light-sensitive Protoporphyrin IX, and activated in the skin by light in the visible spectrum. When skin incubated with 5-ALA subsequently is exposed to light, photoactivated PpIX catalyzes a photochemical reaction, which leads to cell apoptosis of the dysplastic or neoplastic tissue. The amount of PpIX fluorescence in the skin is estimated by PpIX fluorescence measurements on skin surface by fluorescence photographs and in the skin depth with fluorescence microscopy. Previous studies have suggested an association of the amount of PpIX in the skin and the clinical outcome of PDT.

The highly lipophilic nature of the stratum corneum (SC) provides the main barrier for influx of drugs and environmental chemicals into the body (6). SC is the greatest impediment for uptake of 5-ALA and the formation of PpIX can be increased by modifying the SC. Pretreatment of the skin facilitates local uptake of photosensitizing agents and is therefore recommended to obtain optimal outcomes in PDT. Recently, different energy-based devices have been introduced for PDT pretreatment to disrupt the SC barrier and effectively increase PpIX accumulation. However, current light-based treatments, such as ablative and non-ablative lasers, are painful to patients and induce thermal damage that result in oozing, crusting or peeling of the skin.

To increase cutaneous absorption with minimal damage to the skin, thermo-mechanical fractional intervention (TMFI) has been introduced as a new technology. TMFI rapidly transfer thermal energy by a metallic pyramid tip that enable skin contact through integrated pulsed movements. The rapid heating dehydrates the epidermis and superficial dermis and create micropores with no coagulative damage of surrounding tissue. The amount of thermal energy delivered can be adjusted by pulse duration and by the protrusion depth of the tip that sets the thermal matching between the tip and the skin. TMFI has in one study shown to increase uptake of hydrophilic drugs compared with no skin pretreatment. As TMI dehydrates the epidermis, hydrophilic drugs dissolved in a low viscosity liquid-based vehicle may be more readily distributed within the skin compared to drugs dissolved in a high viscosity vehicle.

The investigators hypothesize that i) TMFI increases 5-ALA induced PpIX accumulation compared with no pretreatment and that ii) TMFI + 5-ALA in a low viscosity vehicle formulation enhances PpIX skin biodistribution compared with 5-ALA in a high viscosity vehicle formulation.

Potentially, TMFI pretreatment could improve PpIX biodistribution and reduce photosensitizer incubation time to obtain sufficient PpIX accumulation. This could significantly benefit thousands of patients who each year undergo PDT for dysplastic skin lesions.

ELIGIBILITY:
Inclusion Criteria: Healthy participants above 18 years of age

* Fitzpatrick skin type I-III and normal skin on the upper back
* Fertile women with negative U-hCG and use of safe anticontraceptive during the entire study period e.g. oral hormonal contraceptives, intrauterine devices, subdermal implantation or hormonal vaginal ring
* Provided informed written consent

Exclusion Criteria:

* No previous PDT or laser treatment within the past 6 months in the study areas
* Pregnant or lactating women
* Participants with known allergy to 5-ALA, lidocaine or any excipients to components in the vehicles
* Considered unable to follow the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Change in PpIX fluorescence at skin surface following TMFI and topical 5-ALA in gel and cream vehicle | Baseline and in 30-minute intervals until 3 hours
  Levels of PpIX uptake at the skin surface quantitatively from PpIX imaging.
PpIX fluorescence biodistribution inside skin | 3 hours
  Levels of PpIX uptake inside predefined skin regions: Epidermis, superficial dermis, mid dermis and deep dermis evaluated on fluorescence microscopy images. Biopsies used for fluorescence microscopy was sampled after 3 hours.

SECONDARY OUTCOMES:
Histological skin interactions after TMFI | 3 hours
  Biopsies were stained with haematoxylin and eosin (HE) for light microscopy for histopathology analysis of TMFI effect on the skin. Depth and width of the TMFI effect on the skin was measured.
Severity of local skin reactions | 5 minutes after TMFI pretreatment
  Local skin reaction (LSR)-grading scale. Evaluation of redness, scaling, edema, pustules, and erosion on a 5-point categorial scale of severity. Scores are 0, 1, 2, 3, and 4, for individual parameters:
  Redness: None, slightly pink <50%, pink or light red >50%, red restricted to treatment area, and red extending outside treatment area.
  Scaling: None, isolated scale, scaling <50%, scaling >50%, scaling extending outside treatment area.
  Edema: None, slight specific edema, palpable edema beyond individual lesions, confluent and/or visible edema, and marked swelling extending outside treatment area.
  Pustules: None, vesicles only, transudate or pustules <50%, transudate or pustules >50%, and transudate or pustules extending outside treatment area.
  Erosion: None, lesion specific erosion, erosion extending beyond individual lesion, erosion >50%, and black eschar or ulceration.
Severity of local skin reactions | 3 hours after TMFI pretreatment
  Local skin reaction (LSR)-grading scale. Evaluation of redness, scaling, edema, pustules, and erosion on a 5-point categorial scale of severity. Scores are 0, 1, 2, 3, and 4, for individual parameters:
  Redness: None, slightly pink <50%, pink or light red >50%, red restricted to treatment area, and red extending outside treatment area.
  Scaling: None, isolated scale, scaling <50%, scaling >50%, scaling extending outside treatment area.
  Edema: None, slight specific edema, palpable edema beyond individual lesions, confluent and/or visible edema, and marked swelling extending outside treatment area.
  Pustules: None, vesicles only, transudate or pustules <50%, transudate or pustules >50%, and transudate or pustules extending outside treatment area.
  Erosion: None, lesion specific erosion, erosion extending beyond individual lesion, erosion >50%, and black eschar or ulceration.
Severity of local skin reactions | 14 days after TMFI pretreatment
  Local skin reaction (LSR)-grading scale. Evaluation of redness, scaling, edema, pustules, and erosion on a 5-point categorial scale of severity. Scores are 0, 1, 2, 3, and 4, for individual parameters:
  Redness: None, slightly pink <50%, pink or light red >50%, red restricted to treatment area, and red extending outside treatment area.
  Scaling: None, isolated scale, scaling <50%, scaling >50%, scaling extending outside treatment area.
  Edema: None, slight specific edema, palpable edema beyond individual lesions, confluent and/or visible edema, and marked swelling extending outside treatment area.
  Pustules: None, vesicles only, transudate or pustules <50%, transudate or pustules >50%, and transudate or pustules extending outside treatment area.
  Erosion: None, lesion specific erosion, erosion extending beyond individual lesion, erosion >50%, and black eschar or ulceration.
Presence of perceived pain during treatment | During the actual TMFI pretreatment, estimated 1-2 minute per participant
  VAS Visual analogue scale for perceived pain. Scores are 1, 2, 3, 4, 5, 6, 7, 8, 9, and 10, ranging from none to very severe. Higher is worse, and lower scores for treatment modalities are desirable.
Safety including wounding, scarring, hyper and hypo pigmentation | 14 days
  Safety concerning side-effects evaluated on a 5-point categorial scale for hyper- and hypopigmentation, erosions, and scarring. Scores are 0, 1, 2, 3, and 4, for none, mild, moderate, severe, and very severe. A lower score is desirable.

CONTACTS AND LOCATIONS:
Overall Officials: Merete Hædersdal, DMSc, Study Director — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: No